CLINICAL TRIAL: NCT03996993
Title: Diagnosing and Monitoring Recurrent Disease in Prostate Cancer Patients Using a Positron Emission Tomography Radiotracer (Axumin™)
Brief Title: Defining Recurrent Disease With Axumin™
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Center of Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/12/7
Record Dates: First submitted 2019-06-18; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: prostate cancer; Axumin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; fluciclovine F-18; Leuprolide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Hormone Therapy Cohort: Post-radical prostatectomy patients fitting our inclusion criteria, including rising PSA > 0.1 ng/ml, a positive SOC Axumin scan, and a patients not having received hormonal therapy for a minimum of 3 months, will receive hormonal therapy in the form of Casodex for 2 weeks, followed by Lupron indefinitely. Patients will then receive serial Axumin scans up to 1 year post-therapy.
  Interventions: Drug: Casodex, Axumin
- Salvage Radiotherapy Cohort: Post-radical prostatectomy patients fitting our inclusion criteria, including rising PSA > 0.1 ng/ml, not concurrently on androgen deprivation therapy (ADT) and/or received ADT in the past 3 months, and a positive SOC Axumin scan, will receive salvage radiation therapy according to the following protocol. External beam radiation therapy will be delivered in the form of high-dose intensity modulated radiation therapy (IMRT). A total prescribed dose of 72 Gy will be delivered in 40 fractions over 8 weeks. For the first 25 fractions, the clinical target volume (CTV) is defined as the residual prostatic bed, plus internal/external iliac nodes. For the subsequent 15 fractions the CTV is defined as the residual prostatic bed plus margin. As part of SOC, the radiation fields will incorporate the Axumin positive areas into treatment planning objectives. Patients will then receive serial Axumin scans up to 1 year post-therapy.
  Interventions: Radiation: Salvage Radiation, Axumin

INTERVENTIONS:
Drug: Casodex, Axumin — Patients will receive hormone therapy if Axumin positive area appears.
  Other Names: Lupron
  Groups: Hormone Therapy Cohort
Radiation: Salvage Radiation, Axumin — Patients will receive salvage radiation therapy if Axumin positive area appears.
  Groups: Salvage Radiotherapy Cohort

SUMMARY:
This project seeks to use advanced imaging (specifically, positron emission tomography/computed tomography [PET/CT]) to detect, locate, and characterize recurrent disease in the setting of patients with prostate cancer.

DETAILED DESCRIPTION:
This protocol details the study design for patients with prostate cancer (PCa) who have failed primary treatment with radical prostatectomy, and now have rising PSA as indicated by a recent PSA blood draw value > 0.1 ng/ml. Patients fitting our inclusion criteria for the study, will receive an Axumin scan as part of their standard of care (SOC) treatment. If the SOC scan is positive, patients under this protocol will either subsequently receive hormone therapy OR salvage radiation therapy (not both concurrently). Patient response to therapy will be assessed with serial Axumin scans identifying additional lesions present at 3 months, 6 months, and 12 months (1 year) post-therapy, with the latter time point being our endpoint of the study.

The study aims are as follows:

1. The investigators would like to understand the hormonal therapy response based on Axumin scans administered over a time course of 3 months, 6 months, and 12 months post-hormone therapy treatment.
2. The investigators would like to understand the salvage radiotherapy response based on Axumin scan results incorporated into radiation treatment planning over a time course of 3 months, 6 months, and 12 months post-salvage radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

General requirements:

1. Karnofsky performance status of >50 (or ECOG/WHO equivalent).
2. Age > 18.
3. Ability to understand a written informed consent document, and the willingness to sign it.
4. History of histologically confirmed adenocarcinoma of the prostate and underwent radical prostatectomy for primary treatment with curative intent.
5. Men diagnosed with recurrent/persistent prostate cancer disease following radical prostatectomy based on a detectable or rising PSA value ≥ 0.1 ng/ml.
6. Positive commercial standard of care (SOC) Axumin scan at time of restaging disease.
7. Patients should not have been previously treated for biochemical recurrence (BCR) (i.e., this is the first diagnosis for BCR.
8. Language proficiency in English, Spanish, Japanese, Korean, Vietnamese. Our office has translators to coherently translate the consent documents to patients.

Inclusion criteria specific for patients on response to ADT study:

1. Ability to tolerate androgen deprivation therapy (Casodex and Lupron) indefinitely.
2. Been off ADT for minimum of 3 months.
3. Ability to receive a possible of 4 Axumin PET/CT scans within a year.

Inclusion criteria specific for patients on response to salvage radiotherapy study:

1. Considering salvage radiotherapy.
2. Ability to tolerate salvage radiation therapy for 8 weeks.

Exclusion Criteria:

General requirements:

1. Patients not capable of getting PET study due to weight, claustrophobia, allergic reaction, and/or inability to lay still for the duration of the exam.
2. Women and children.
3. Men currently on or seeking primary treatment (surgery or radiation) for prostate cancer.
4. History of bilateral orchidectomy.
5. Neoadjuvant chemotherapy or radiation therapy prior to prostatectomy. This includes focal ablation techniques (HiFu).
6. Ongoing treatment with any systemic therapy intended for the treatment of prostate cancer (e.g., antiandrogen or LHRH agonist or antagonist).
7. Prior history of any other malignancy within the last 2 years, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer.

Exclusion criteria specific for patients on response to ADT study:

1. Being considered for salvage radiotherapy.
2. Androgen deprivation therapy (ADT) in the past 3 months.

Exclusion criteria specific for patients on response to salvage radiotherapy study:

1. Currently on ADT or on ADT within the past 3 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men with recurrent prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of baseline Axumin uptake | 2019-2020
  Utilizing standard uptake values (SUV) from the tumor origin, serial Axumin SUV values will be calculated as a percentage of the baseline SUV value.

SECONDARY OUTCOMES:
PSA blood draw | 2019-2020
  Prostate specific antigen (PSA) values expressed as [ng/ml] will be serially drawn at each time of the Axumin scan to correlate with percentage of baseline SUV value.

CONTACTS AND LOCATIONS:
Locations (1):
- Kenneth Tokita, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Undecided